CLINICAL TRIAL: NCT03669796
Title: A Study of the Effects of Marine Protein Hydrolysate as Dietary Supplement on the Regulation of Postprandial Blood Glucose Metabolism in Healthy Subjects
Brief Title: Marine Protein Hydrolysate as Dietary Supplement in Elderly Part I
Acronym: MPH-BS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017/1794
Record Dates: First submitted 2018-07-02; First posted 2018-09-13 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
Keywords: Dietary Supplements; Fish Proteins; Protein Hydrolysates; Aged
MeSH Terms: interventions — 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Intervention Model Description: A double-blind crossover trial, including two different study days, with 4-7 days wash-out (WO) period in between. The intervention implemented 20 mg of MPH per kg body weight (test material) or control (casein).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supplementary Marine protein hydrolysate (Experimental): 20 mg powder per kg body weight of Marine protein hydrolysate (MPH)
  Interventions: Dietary Supplement: Marine protein hydrolysate (mph)
- control (Placebo Comparator): 20 mg powder per kg body weight of casein/maltodextrin
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Marine protein hydrolysate (mph) — Marine (Cod) protein hydrolysate
  Arms: supplementary Marine protein hydrolysate
Dietary Supplement: Control — Maltodextrin/Casein
  Arms: control

SUMMARY:
The aim of this study is to investigate the potential effect of a marine protein hydrolysate (MPH) supplement before a meal on postprandial glucose tolerance in healthy subjects, to achieve more knowledge on this presumed beneficial, blood glucose lowering effect

DETAILED DESCRIPTION:
To further investigate the effects of MPH in a single dose of 20 mg/kg of body weight on postprandial blood glucose, insulin and GLP-1 (as markers of glucose metabolism) in healthy, active middle-aged to elderly subjects - age 40-65 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Body mass index (BMI) 20-30

Exclusion Criteria:

* Suspected allergies against fish or shellfish
* Low or unstable blood pressure
* Diabetes mellitus, treated pharmacological
* Chronic diseases or therapies that is likely to interfere with the evaluation of study results
* Acute infections (may be reconsidered for inclusion at a later time)
* Allergic to milk, confirmed diagnose
* Pregnancy
* Women who are breast-feeding infants
* Inability or unwillingness to comply with the requirements of study procedures

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Glucose | First sample fasting baseline, thereafter repeated samples every 20 minutes (i.e.20, 40, 60, 80, 100,120,140 minutes after baseline), last at 200 minutes after baseline.
  Postprandial glucose (mmol/L) change on each day of intervention

SECONDARY OUTCOMES:
Insulin | First sample fasting baseline, thereafter repeated samples every 20 minutes (i.e.20, 40, 60, 80, 100,120,140 minutes after baseline), last at 200 minutes after baseline
  Postprandial Insulin (mIE/L) - change on each day of intervention
Hormon 1 | First sample fasting baseline, thereafter repeated samples (i.e.20, 40, 60, 100 minutes after baseline), last at 200 minutes after baseline
  Glucagon like peptide 1 (GLP-1) pmol/l change on each day of intervention
Visual analogue scale (VAS) | First (baseline) symptomscore (as described above) measured fasting , thereafter repeated symptom score i.e. at 20, 40 minutes after baseline, last symptom score measure at 200 minutes after baseline
  Assessed by questionnaire VAS, scale from 0-10, where 0 is minimum score and 10 is the maximum score, reported e.g. as a total score of 7. The higher the reported value is the worse outcome.
KANE, symptom score | First (baseline) symptom score (as described above) measured fasting and the next measure at 200 minutes after baseline
  Assessed by questionaire KANE (family name) , scale from 0-10, where 0 is minimum score and 10 is the maximum score, reported e.g. as a total score of 7. The higher the reported value is the worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dag Arne Lihaug Hoff, MD, PhD, Study Director — Møre & Romsdal Hospital Trust, Ålesund Hospital
Locations (2):
- Norway (2):
  - Ålesund Hospital, Helse Møre og Romsdal HF, Ålesund
  - Haukeland University Hospital, Bergen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dale HF, Jensen C, Hausken T, Lied E, Hatlebakk JG, Bronstad I, Lihaug Hoff DA, Lied GA. Effect of a cod protein hydrolysate on postprandial glucose metabolism in healthy subjects: a double-blind cross-over trial. J Nutr Sci. 2018 Nov 28;7:e33. doi: 10.1017/jns.2018.23. eCollection 2018. PMID 30524707
- [Result] Dale HF, Jensen C, Hausken T, Lied E, Hatlebakk JG, Bronstad I, Hoff DAL, Lied GA. Erratum: Effect of a cod protein hydrolysate on postprandial glucose metabolism in healthy subjects: a double-blind cross-over trial - CORRIGENDUM. J Nutr Sci. 2019 Jan 18;8:e1. doi: 10.1017/jns.2018.30. eCollection 2019. PMID 30719283
- [Result] Dale HF, Jensen C, Hausken T, Lied E, Hatlebakk JG, Bronstad I, Hoff DAL, Lied GA. Acute effect of a cod protein hydrolysate on postprandial acylated ghrelin concentration and sensations associated with appetite in healthy subjects: a double-blind crossover trial. Food Nutr Res. 2019 Oct 22;63. doi: 10.29219/fnr.v63.3507. eCollection 2019. PMID 31692759